CLINICAL TRIAL: NCT01783262
Title: The Role of Extracorporeal Shock Wave Therapy in the Treatment of Trapezial-Metacarpal Osteoarthritis.
Brief Title: The Role of Extracorporeal Shock Wave Therapy in the Treatment of Trapezial-Metacarpal Osteoarthritis. A Double Blind Randomized Controlled Study.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Francesco Ioppolo, MD, PhD, University of Roma La Sapienza
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: Interventional Study Design
Record Dates: First submitted 2013-01-29; First posted 2013-02-04 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Osteoarthritis Trapezial-metacarpal Joint

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extracorporeal shock wave therapy (Active Comparator): an energy level of 0.09 mJ/mm2, 2400 pulses once a week for 4 weeks.
  Interventions: Device: Extracorporeal shock wave therapy STORZ MEDICAL Modulith SLK
- sham extracorporeal shock wave therapy (Placebo Comparator): The second grouop of patients received 0.04 mJ/mm2, 2400 pulses once a week for 4 weeks.
  Interventions: Device: Device: Sham extracorporeal shock wave therapy STORZ MEDICAL Modulith SLK

INTERVENTIONS:
Device: Extracorporeal shock wave therapy STORZ MEDICAL Modulith SLK — an energy level of 0.09 mJ/mm2, 2400 pulses once a week for 4 weeks.
  Arms: Extracorporeal shock wave therapy
Device: Device: Sham extracorporeal shock wave therapy STORZ MEDICAL Modulith SLK
  Other Names: an energy level of 0.09 mJ/mm2, 2400 pulses once a week for 4 weeks.
  Arms: sham extracorporeal shock wave therapy

SUMMARY:
Evaluate if extracorporeal shock wave therapy is more effective than sham treatment in patients with trapezial-metacarpal osteoarthritis in pain relief and functional improvement.

ELIGIBILITY:
Inclusion Criteria:

* according to the Eaton et al. classification the inclusion criteria involved those patients with stage III, participants had to have a history 6 months of pain and they were 18 years of age or older. Exclusion criteria were also the presence of degenerative or non-degenerative neurologic conditions, in which pain perception is altered, a history of coagulopathy, cancer, cardiac pacemaker, calcaneal fracture, and pregnancy.

Exclusion Criteria:

* Exclusion criteria were also the presence of degenerative or non-degenerative neurologic conditions, in which pain perception is altered, a history of coagulopathy, cancer, cardiac pacemaker, calcaneal fracture, and pregnancy.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2009-12; Primary Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale | The change in the mean Visual Analogic Scale scores from baseline to 3 and 6 months after the intervention
  It is a horizontal line, 10 cm in length with 0 cm labeled "no pain" and 10 cm labeled "worst pain I have ever had". The patient marks on the line the point that they feel represents their perception of their current state
Duruöz Hand Index (DHI) | The change in the mean of DHI at 3 and 6 months follow up
  is a self-report questionnaire which measures hand functional ability detecting how much difficulty the patient has performing eighteen daily tasks of living in reference to hand function. Each item is scored from 0 (performed without difficulty) to 5 (impossible to do). A total score is obtained by adding the scores of all questions (range 0-90). A higher score indicates greater disability. It was found that this scale is reliable and valid in patients with osteoarthritis
Disabilities of the Arm, Shoulder, and Hand questionnaire | The changes in mean at 3 and 6 months follow up
  It is a 30-item scale that addresses difﬁculty in performing various physical activities that require upper extremity function (physical function, 21 items); symptoms of pain, activity-related pain, tingling, weakness, and stiffness (pain symptoms, 5 items); or impact of disability and symptoms on social activities, work, sleep, and psychological well-being (emotional and social function, 4 items). The score ranges from 0 to 100, where 0 disability and 100 most severe disability.

SECONDARY OUTCOMES:
grip and pinch tests | The change in mean at 3 and 6 months follow up
  The measure of strength by hand grip and pinch tests, for continuous variables that were measured in kilograms with a standard dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- La Sapienza University, Rome, Italy, Italy